CLINICAL TRIAL: NCT05956665
Title: Adapting the Shed-MEDS Deprescribing Intervention to Dementia Care in Assisted Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer Kim, Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: #230560
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Polypharmacy; Dementia; Quality of Life
Keywords: Deprescribing
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: All participants will receive a clinical review of their prescribed medications by a research clinician, followed by a resident/surrogate interview to assess their willingness to discontinue or reduce some of their medicines based on the clinical recommendations of the research clinician. The facility's medical providers will also be part of the deprescribing decision process and will initiate any agreed upon deprescribing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ShedMEDS Intervention (Experimental): ShedMEDS is a patient-centered intervention to safely deprescribe medicines, as defined by dose reductions and stopping, based on a combination of clinical criteria and patient/surrogate preference.
  All participants received a clinical review of their medications by a research nurse practitioner, followed by a resident/surrogate interview to assess their willingness to discontinue or reduce some of their medicines based on the research clinician's clinical recommendations. The deprescribing recommendations were discussed with the assisted living facility's medical providers, who initiated the agreed upon deprescribing.
  Interventions: Behavioral: Shed-MEDS deprescribing intervention

INTERVENTIONS:
Behavioral: Shed-MEDS deprescribing intervention — See single arm description

SUMMARY:
This single-arm pilot study will evaluate the effects of an intervention to reduce exposure to unnecessary or potentially harmful medications among residents with dementia living in an assisted living facility. The goal of the intervention is to safely deprescribe medications (defined by dose reductions and stopped medications), based on a combination of clinical criteria and resident/surrogate preferences. The investigators will evaluate the effects of the intervention on the total number of medications deprescribed from enrollment at 30, 60, and 90 days along with resident/surrogate reports of quality of life at enrollment and 90 days.

DETAILED DESCRIPTION:
This single-arm pilot trial will evaluate an evidence-based, patient-centered deprescribing intervention with assisted living facility (ALF) residents age 65+ who have a diagnosis of dementia. This deprescribing intervention was demonstrated to be safe and effective in reducing medication burden during the Shed-MEDS randomized clinical trial that enrolled hospitalized older adults discharging to post-acute care facilities. The intervention includes a comprehensive review of a participant's medications by the study's clinician and deprescribing recommendations using evidence-based guidelines. Deprescribing recommendations will be shared with residents/surrogate decision makers (i.e., respective family member/s) to determine their willingness to stop or reduce the dose of the targeted medications. If the resident/surrogate-decision maker agrees, deprescribing recommendations will then be communicated with the routine ALF medical providers for consideration and final deprescribing decisions.

ELIGIBILITY:
Inclusion Criteria:

* Resident of assisted living facility
* Speaks English (due to interview-based assessments)
* Diagnosis of dementia
* Taking a total of 5 medications or at least one potentially inappropriate medication (defined by the Beers criteria, STOPP criteria, and the Rationalization of home medication by an Adjusted STOPP in older Patients [RASP])
* Able self-consent or has a proxy (surrogate)

Exclusion Criteria:

- None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Abe's Garden Community, Nashville, Tennessee
  - NHC At The Trace, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared, per written request, upon study completion and all final analyses

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from memory care units at two assisted living facilities in Nashville, TN.
Groups:
- ShedMEDS Intervention: ShedMEDS is a patient-centered intervention to safely deprescribe medicines, as defined by dose reductions and stopping, based on a combination of clinical criteria and patient/surrogate preference.
  All participants received a clinical review of their medications by a research nurse practitioner, followed by a resident/surrogate interview to assess their willingness to discontinue or reduce some of their medicines based on the research clinician's clinical recommendations. The deprescribing recommendations were discussed with the assisted living facility's medical providers, who initiated the agreed upon deprescribing.
  Shed-MEDS deprescribing intervention: See single arm description
Period: Overall Study
Arm/Group | ShedMEDS Intervention
Started | 18
Intervention | 16
30-Day Follow Up | 16
60-Day Follow Up | 16
Completed | 16
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One participant withdrew consent prior to completing baseline data collection and is therefore excluded from the analysis.
Arm/Group | ShedMEDS Intervention
Number analyzed (Participants) | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 82 [77.5 to 87.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Brief Interview for Mental Status (BIMS) [Median (Inter-Quartile Range); unit: units on a scale] — The BIMS is a standardized assessment to screen for cognitive impairment with a score range of 0-15. A total score of 0-7 represents severe impairment, 8-12 moderate impairment, and 13-15 cognitively intact.
  units on a scale | 2.5 [0.3 to 6.8]
Charlson Comorbidity Index (CCI) [Median (Inter-Quartile Range); unit: units on a scale] — The Charlson Comorbidity Index is calculated by summing the weights of all comorbid conditions documented in the participant's medical record. There is an additional 1 point increase in score for every decade starting at age 50. The age adjusted score ranges from 0-31 with higher scores indicating more comorbid illness.
  units on a scale | 5.0 [5.0 to 6.5]
Total Number of Medications [Median (Inter-Quartile Range); unit: Medications] — The number of medications a participant takes. This includes all prescribed and over-the-counter medications and both scheduled and as-needed (PRN) medications.
  Medications | 13 [8 to 15]
Anticholinergic & Sedative Drug Burden Index [Median (Inter-Quartile Range); unit: units on a scale] — A Drug Burden Index (DBI) score is calculated for each anticholinergic and sedative medication by dividing the individual medication's prescribed daily dose by the sum of the minimum effective dose (per FDA minimum recommended dose) and the patient's daily dose. The score range for each individual medication is 0 to 1, and the Anticholinergic & Sedative DBI reported is the sum of the individual medication scores. The Anticholinergic & Sedative DBI has a minimum score of 0 and no maximum. Higher scores indicate a higher drug burden (i.e., lower score is a better outcome).
  units on a scale | 2.3 [0.9 to 3.7]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Medications That Have Been Deprescribed Since Enrollment
Description: The number of medications (including all prescribed and over-the-counter medications and both scheduled and as-needed medications) that have been deprescribed since enrollment. Deprescribed is defined as either stopping or reducing the dose/frequency of a medication.
Time Frame: 30 days
Population: All participants who completed the intervention protocol (medication review, surrogate interview, and provider conversation).
Measure: Median (Inter-Quartile Range); unit: Medications
Arm/Group | ShedMEDS Intervention
Number analyzed (Participants) | 16
Medications | 4 [2.25 to 6.00]

2. Primary Outcome: Total Number of Medications That Have Been Deprescribed Since Enrollment
Description: as for outcome 1
Time Frame: 60 days
Population: All participants who completed and the entire intervention protocol (medication review, surrogate interview, and provider conversation).
Measure: Median (Inter-Quartile Range); unit: Medications
Arm/Group | ShedMEDS Intervention
Number analyzed (Participants) | 16
Medications | 4 [2.25 to 6.75]

3. Primary Outcome: Total Number of Medications That Have Been Deprescribed Since Enrollment
Description: as for outcome 1
Time Frame: 90 days
Population: All participants who completed the entire intervention protocol (medication review, surrogate interview, and provider conversation).
Measure: Median (Inter-Quartile Range); unit: Medications
Arm/Group | ShedMEDS Intervention
Number analyzed (Participants) | 16
Medications | 4 [2.25 to 7.00]

4. Primary Outcome: Resident Quality of Life
Description: The Dementia Quality of Life Instrument-Proxy Version (DEMQOL-Proxy) is used to evaluate health-related quality of life in participants with severe dementia as rated by their caregivers. The DEMQOL-Proxy has 31 items which are reported on a four-point Likert scale (a lot/ quite a bit/ a little/ not at all) with a total score range from 31 to 124. Higher scores indicate a better health-related quality of life (i.e., higher scores are better).
Time Frame: Enrollment
Population: All participants who completed the entire intervention protocol
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ShedMEDS Intervention
Number analyzed (Participants) | 16
score on a scale | 94 [85.5 to 106.5]

5. Primary Outcome: Resident Quality of Life
Description: as for outcome 4
Time Frame: 90 days
Population: All participants who completed the intervention protocol
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ShedMEDS Intervention
Number analyzed (Participants) | 16
score on a scale | 104.5 [95.3 to 109.5]

ADVERSE EVENTS:
Time Frame: All adverse events including serious adverse events and all-cause mortality were continuously monitored from participant enrollment through final follow-up 90-days after intervention completion.
Description: The study used NIH/NIA definition for adverse and serious adverse events. Serious adverse events included hospitalization and death. Non-serious adverse events were defined as emergency room visits, which did not lead to a subsequent hospitalization. Data for all unplanned healthcare utilization and death are reported here regardless of cause or study-relatedness.
Arm/Group | ShedMEDS Intervention
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShedMEDS Intervention (N=18)
Heart Failure (Cardiac disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShedMEDS Intervention (N=18)
Fall (Injury, poisoning and procedural complications) | 5 (5)
Mental Status Change (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT05956665/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT05956665/ICF_001.pdf